CLINICAL TRIAL: NCT01402102
Title: Efficacy and Safety of Aged Garlic Powder on Lipids
Brief Title: A Human Trial to Evaluate the Efficacy and Safety of Aged Garlic Powder on Improvement of Blood Lipids in Subjects With Hyperlipidemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Doul-BGarlic-001
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Results first posted 2012-10-04 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Hyperlipidemia
Keywords: Aged garlic; Hyperlipidemic; LDL; HDL; Triglyceride
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aged garlic powder (Experimental)
  Interventions: Dietary Supplement: Aged garlic powder
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo powder

INTERVENTIONS:
Dietary Supplement: Aged garlic powder — Aged garlic powder(6.0g/day)
  Arms: Aged garlic powder
Dietary Supplement: Placebo powder — Placebo powder(6.0g/day)
  Arms: Placebo

SUMMARY:
We performed a double-blind parallel study in a group of mildly hypercholesterolemic subjects who were given aged garlic powder over a period of 12 weeks. We measured serum lipids, including total cholesterol, low-density-lipoprotein (LDL) and high-density-lipoprotein (HDL) cholesterol, and triglycerides, and monitored their blood pressure.

DETAILED DESCRIPTION:
An increased serum cholesterol level is an important risk factor for the development of cardiovascular and cerebrovascular disease. Reduction of these and other risk factors through dietary modification, behavioral changes, and medicinal intervention has already substantially decreased the incidence and mortality from cardiovascular and cerebrovascular disease. Supplementation of the diet with certain biofactors may further reduce such risk factors. Aged garlic belongs to a group of dietary supplements that may lessen the incidence of cardiovascular and cerebrovascular disease by reducing lipids levels and decreasing platelet responsiveness to activating agents.

ELIGIBILITY:
Inclusion Criteria:

* Mild hypercholesterolemic subjects aged from 20 to 80 years
* had no received lipid-lowering drugs for at least 3 months prior to the recruitment

Exclusion Criteria:

* self-reported pregnancy,lactation
* prevalent heart disease,cancer,renal disorder, or diabetes mellitus, and use of lipid or antihypertensive medications

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dal-Sik Kim, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 20 to 80 years, a BMI(Body Mass Index)>23 kg/m^2, an LDL-C(Low Density Lipoprotein-cholesterol) concentration between 130 and 220 mg/dL. Subjects were excluded if they had heart disease, liver or kidney disease, irregular lifestyle habits, or if they took medication and functional foods known to affect lipid metabolism
Groups:
- Aged Garlic Powder: Oral intake Aged garlic powder(6.0g/day) for 12weeks.
- Placebo: Oral intake placebo(6.0g/day) for 12weeks
Period: Overall Study
Arm/Group | Aged Garlic Powder | Placebo
Started | 30 | 30
Completed | 28 | 27
Not Completed | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Insufficiency of compliance | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aged Garlic Powder | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 46
  >=65 years | 8 | 6 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.2) | 50.8 (8) | 50.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 12 | 8 | 20
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Changes in LDL-cholesterol(Low Density Lipoprotein - Cholesterol)
Description: LDL-C(Low Density Lipoprotein - cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
mg/dl
  Pre | 150.6 (14.1) | 150.1 (15.7)
  Post | 155.8 (21.9) | 156.3 (29.8)

2. Secondary Outcome: Changes in HDL-Cholesterol(High Density Lipoprotein - Cholesterol)
Description: HDL-cholesterol(High Density Lipoprotein - cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: PP analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Aged Garlic Powder: Aged garlic powder 6.0g/day oral intake
- Placebo: Placebo 6.0g/day oral intake
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
mg/dl
  Pre | 46.86 (9.40) | 50.81 (9.19)
  Post | 50.36 (8.85) | 50.48 (9.76)

3. Secondary Outcome: Changes in Triglycerides
Description: Triglyceride was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: PP analysis
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
mg/dl
  Pre | 139.79 (54.55) | 124.11 (47.65)
  Post | 120.21 (63.61) | 128.11 (65.50)

4. Secondary Outcome: Changes in Total Cholesterol
Description: Total cholesterol was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
mg/dL
  Pre | 241.07 (23.97) | 228.93 (20.01)
  Post | 233.50 (24.63) | 227.33 (32.51)

5. Secondary Outcome: Changes in Apo-A1(Apolipoprotein A1)
Description: Apo-A1(Apolipoprotein A1) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
g/L
  Pre | 1.48 (0.21) | 1.43 (0.18)
  Post | 1.41 (0.19) | 1.39 (0.17)

6. Secondary Outcome: Changes in Apo-B(Apolipoprotein B)
Description: Apo-B(Apolipoprotein B) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
g/L
  Pre | 1.21 (0.13) | 1.03 (0.14)
  Post | 1.07 (0.12) | 1.01 (0.19)

7. Secondary Outcome: Changes in FFA(Free Fatty Acid)
Description: FFA(free fatty acid) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12 weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: µEq/L
Arm/Group | Aged Garlic Powder | Placebo
Number analyzed (Participants) | 28 | 27
µEq/L
  Pre | 570.25 (193.02) | 554.04 (179.64)
  Post | 618.14 (184.78) | 523.93 (222.93)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Aged Garlic Powder | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No